CLINICAL TRIAL: NCT05322044
Title: Financial Incentives to Improve Adherence to Inhaled Asthma Medications in Children and Young People With Asthma
Brief Title: Financial Incentives to Improve Asthma
Acronym: FINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22SM7433; 306829 (Other: IRAS)
Record Dates: First submitted 2022-03-16; First posted 2022-04-11 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Asthma in Children; Medication Adherence
Keywords: Electronic monitoring device; Financial incentives; Reminders; Asthma control
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (no financial incentive) (No Intervention): No incentive. Usual care (plus EMD with reminders) for 12-weeks.
- Intervention (financial incentive) (Experimental): Financial incentive dependent upon daily medication adherence (plus EMD with reminders) for 12-weeks.
  Interventions: Behavioral: Financial incentives

INTERVENTIONS:
Behavioral: Financial incentives — Financial incentives dependent upon adherence will be given to participants alongside additional EMD associated app features for 12-weeks.
  Arms: Intervention (financial incentive)

SUMMARY:
The aim of this pilot randomised controlled trial is to assess the effectiveness of a short-term financial incentives intervention at bringing about behaviour change, namely short-medium term improvements in inhaled corticosteroid (ICS) adherence and asthma control in children and young people (CYP) with asthma.

DETAILED DESCRIPTION:
After obtaining informed consent from parents (and assent from the CYP), CYP will be enrolled in a 24-week programme. All participants will receive an electronic monitoring device (EMD) which will be programmed with twice daily audio-visual reminders and will be required to download the EMD-associated App onto their smartphones. All participants will be required to attend 3 study visits at 0 weeks (baseline), 12-weeks and 24-weeks (follow-up).

At baseline participants will be assessed for inhaler technique and given an asthma action plan (if they do not have one already) and will be randomised to either the control group or the intervention group. Intervention period will run between study visit 1 (0-weeks) and study visit 2 (12-weeks). Over the intervention period, participants in the intervention group will use their EMD with reminders, but will also be given financial incentives dependent upon their daily adherence and will have access to some additional EMD-associated app features (including notifications, a reward totaliser and a traffic light calendar to monitor progress). Control group participants will receive their usual care plus the use of EMD with reminders over the intervention period.

After the intervention period (at study visit 2), intervention participants will no longer receive rewards or be able to access the additional app features. All participants (control and intervention) will be able to use their EMD with reminders for the final 12-week follow-up period.

After completion of the 24-week programme, all participants will be required to return their EMD devices and will be invited to a focus group to share experiences and feedback of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from parent/guardian and assent from child.
* CYP with doctor diagnosed asthma presenting to Emergency Department (ED) with a severe asthma exacerbation (as defined by ERS/ATS guidelines).
* Aged between 11 and 17 years old
* Prescribed maintenance inhaled corticosteroids (ICS) (which can include maintenance and reliever therapy MART) for at least 6-months.
* Own their own mobile smartphone (running Android 8 or higher, or iOS 13 or higher)
* Prescribed the following inhalers: Clenil, Flixotide, Symbicort, Seretide

Exclusion Criteria:

* Parent/guardian / CYP unable to provide consent / assent
* CYP with other, co-existing respiratory conditions
* Parent/guardian/CYP who are not fluent or able to understand the information provided in English.
* CYP who are involved in other intervention research studies (including CTIMPs)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Maconochie, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Started | 16 | 16
Completed | 12 | 13
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.31 (1.58) | 13.50 (1.75) | 13.4 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 10 | 11 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 2 | 5
  Mixed, Mulitple ethnic groups | 4 | 3 | 7
  Asian or Asian British | 2 | 4 | 6
  Black, African, Caribbean, or Black British | 5 | 5 | 10
  Other ethnic group | 2 | 2 | 4
Time since ED presentation [Median (Full Range); unit: days] | 35.5 [16 to 92] | 41 [14 to 139] | 41 [14 to 139]
English primary language at home [Count of Participants; unit: Participants] | 11 | 14 | 25
Asthma Control Test (ACT) [Median (Full Range); unit: units on a scale] — Asthma Control Test (ACT) is a questionnaire measuring asthma control over the past 4-weeks. It consists of 5 questions, each of which are scored using a 5 point Likert scale. A total score is calculated; the minimum possible score is 5 and maximum possible score is 25; a score of 19 and below indicates poor asthma control.
  units on a scale | 20.5 [12 to 25] | 20 [10 to 25] | 20 [10 to 25]
Maintenance asthma treatment [Count of Participants; unit: Participants]
  Clenil modulite | 4 | 11 | 15
  Symbicort Turbohaler | 6 | 4 | 10
  Seretide Evohaler | 6 | 1 | 7
Maintenance asthma treatment step [Count of Participants; unit: Participants]
  Combination (ICS/LABA) | 12 | 5 | 17
  ICS-only | 4 | 11 | 15
Maintenance and Reliever Treatment (MART) regime [Count of Participants; unit: Participants] | 0 | 3 | 3
Multiple daily asthma medications [Count of Participants; unit: Participants]
  Asthma maintenance treatment alone | 8 | 12 | 20
  + 1 other medication | 5 | 3 | 8
  + 2 other medication | 3 | 0 | 3
  + 3 other medication | 0 | 1 | 1
Medication Adherence Reporting Scale for Asthma (MARS-A) [Median (Full Range); unit: units on a scale] — Medication Adherence Reporting Scale for Asthma (MARS-A) is a measure of maintenance treatment adherence. It consists of 10 questions, each question is scored using a Likert scale of 1-5. An average score from all questions is calculated. A minimum possible score is 1 and a maximum score is 5; a score of 4.5 and above indicates high levels of maintenance treatment adherence.
  units on a scale | 4.20 [2.90 to 4.70] | 4.10 [2.60 to 4.70] | 4.20 [2.60 to 4.70]
Illness perceptions (Brief Illness Perceptions Questionnaire, B-IPQ) [Median (Full Range); unit: units on a scale] — Brief Illness Perceptions Questionnaire (B-IPQ) is a measure of illness perceptions. It consists of 8 questions, each question is score on a scale of 0-10 and overall score is calculated. Minimum score is 0 and maximum score is 80. Those with a higher overall score perceive their illness as more threatening.
  units on a scale | 26 [6 to 46] | 33 [12 to 49] | 32 [6 to 49]
Habit (Self Report Behavioural Automaticity Index, SRBAI) [Mean (Standard Deviation); unit: units on a scale] — Self-Report Behavioural Automaticity Index (SRBAI) is a measure of habit. It consists of 4 questions, each question is scored using a Likert scale of 1-5. The average of all questions is calculated, minimum score of 1 and maximum score of 5 and higher scores indicate stronger habit.
  units on a scale | 2.75 (1.09) | 2.91 (0.63) | 2.83 (0.88)
Beliefs in Medicine (BMQ) - Necessity [Mean (Standard Deviation); unit: units on a scale] — Belief in Medicines Questionnaire (BMQ) is a questionnaire to measure beliefs about medicines. It consists of 18 questions, each question is scores using a Likert scale of 1-5. The BMQ is interpreted in 4 sub-sets. 'Necessity' is a sub-set which is calculated from total of questions 1-5 (minimum score 5, maximum score 25), a higher score indicates high levels of belief in the need for medicines.
  units on a scale | 15.19 (3.33) | 14.19 (3.25) | 14.69 (3.28)
Beliefs in Medicine (BMQ) - Concerns [Mean (Standard Deviation); unit: units on a scale] — Belief in Medicines Questionnaire (BMQ) is a questionnaire to measure beliefs about medicines. It consists of 18 questions, each question is scores using a Likert scale of 1-5. The BMQ is interpreted in 4 sub-sets. 'Concerns' is a sub-set which is calculated from total of questions 6-10 (minimum score 5, maximum score 25), a higher score indicates high levels of belief in concern of medicines.
  units on a scale | 15.63 (2.33) | 14.31 (3.42) | 14.97 (2.96)
Beliefs in Medicine (BMQ) - Harm [Median (Full Range); unit: units on a scale] — Belief in Medicines Questionnaire (BMQ) is a questionnaire to measure beliefs about medicines. It consists of 18 questions, each question is scores using a Likert scale of 1-5. The BMQ is interpreted in 4 sub-sets. 'Harm' is a sub-set which is calculated from an average of questions 11-14 (minimum score 4, maximum score 20), a higher score indicates high levels of belief in the harm for medicines.
  units on a scale | 12.5 [6 to 17] | 12 [9 to 20] | 12 [6 to 20]
Beliefs in Medicine (BMQ) - Overuse [Median (Full Range); unit: units on a scale] — Belief in Medicines Questionnaire (BMQ) is a questionnaire to measure beliefs about medicines. It consists of 18 questions, each question is scores using a Likert scale of 1-5. The BMQ is interpreted in 4 sub-sets. 'Overuse' is a sub-set which is calculated from total of questions 15-18 (minimum score 4, maximum 20), a higher score indicates high levels of belief in the overuse of medicines.
  units on a scale | 15 [10 to 17] | 15 [10 to 18] | 15 [10 to 18]
Motivation (adapted Treatment Self-Regulation Questionnaire, TSRQ) - autonomous [Median (Full Range); unit: units on a scale] — Treatment Self-Regulation Questionnaire (TSRQ) was adapted for this study to measure autonomous and controlled motivation. It consists of 8 questions, each question is scored using a Likert scale of 1-7. Autonomous motivation is measured from 4 questions and controlled motivation is measured from the other 4 questions; a total score is calculated with a minimum of 4 and a maximum of 28. The motivation component with the highest total score (e.g., autonomous or controlled) reflects whether an individual is more motivated by external or internal sources.
  units on a scale | 22.50 [8 to 28] | 22.50 [13 to 28] | 22.50 [8 to 28]
Motivation (adapted Treatment Self-Regulation Questionnaire, TSRQ) - controlled [Mean (Standard Deviation); unit: units on a scale] — Treatment Self-Regulation Questionnaire (TSRQ) was adapted for this study to measure autonomous and controlled motivation. It consists of 8 questions, each question is scored using a Likert scale of 1-7. Autonomous motivation is measured from 4 questions and controlled motivation is measured from the other 4 questions; a total score is calculated with a minimum of 4 and a maximum of 28. The motivation component with the highest total score (e.g., autonomous or controlled) reflects whether an individual is more motivated by external or internal sources.
  units on a scale | 18.19 (5.39) | 16.81 (5.08) | 17.50 (5.20)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Percentage ICS Adherence Between Groups at 12-weeks
Description: Comparison of average % ICS adherence measured by EMD for intervention group participants and average % ICS adherence measured by EMD for control group participants at 12-weeks (post-intervention period). EMD will electronically record date/time of asthma inhaler actuation. Data from EMD will be downloaded at study visit/s. Possible scores: 0% (poor adherence) to 100% (good adherence).
Time Frame: Comparison between groups at study visit 2 (12-weeks)
Measure: Median (Full Range); unit: percentage adherence
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 13 | 11
percentage adherence | 56 [7 to 87] | 73 [23 to 89]

2. Secondary Outcome: Proportion of Participants Achieving Good Asthma Adherence (≥80%)
Description: The proportion of participants is defined as number of participants achieving an average % ICS adherence measured by EMD of 80% and above from each group (intervention or control)bat study visit 2 and study visit 3. Within and between group comparisons between groups will be explored.
Time Frame: study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Number; unit: participants
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 13 | 11
participants
  12-weeks | 1 | 4
  24-weeks: number analyzed (Participants) | 12 | 8
  24-weeks | 0 | 0

3. Secondary Outcome: Number of Asthma Exacerbation Needing a Course of Oral Corticosteroids (OCS)
Description: Numbers of asthma exacerbations will be recorded by self-report from parents/child at study visit 2 and 3. Within and between group comparisons between groups will be explored.
Time Frame: study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Number of participants decreased between 12- and 24-weeks due to participant withdrawal
Measure: Count of Participants; unit: Participants
Groups:
- Control (no Financial Incentives): No incentive. Usual care (plus EMD with reminders) for 12-weeks
- Intervention (Financial Incentives): Financial incentive dependent upon daily medication adherence (plus EMD with reminders) for 12-weeks.
  Financial incentives: Financial incentives dependent upon adherence will be given to participants alongside additional EMD associated app features for 12-weeks.
Arm/Group | Control (no Financial Incentives) | Intervention (Financial Incentives)
Number analyzed (Participants) | 14 | 15
Participants
  12-weeks | 1 | 2
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 0 | 1

4. Secondary Outcome: Asthma Control
Description: Measured by validated, self-report Asthma Control Test (ACT). Minimum score of 0 - maximum score of 25. Higher scores = well controlled asthma. Within and between group comparisons between groups will be explored at all study visits.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 20.50 [12 to 25] | 20.00 [10 to 25]
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 21.00 [13 to 25] | 23.00 [11 to 25]
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 22.50 [14 to 25] | 24.00 [17 to 25]

5. Secondary Outcome: Exhaled Nitric Oxide
Description: Measured by FENO which measures nitric oxide level in parts per billion (PPB) in the air you slowly exhale out of child's lungs to be completed by child at each study visit. For children, <20 ppb is low/normal and >35ppb is high. Within and between group comparisons between groups will be explored.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: ppb
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 15 | 16
ppb
  0-weeks | 24 [5 to 122] | 51 [7 to 300]
  12-weeks: number analyzed (Participants) | 10 | 10
  12-weeks | 55.50 [8 to 145] | 66.50 [23 to 205]
  24-weeks: number analyzed (Participants) | 6 | 4
  24-weeks | 46.50 [11 to 56] | 102 [87 to 121]

6. Secondary Outcome: Brief Illness Perceptions Questionnaire (B-IPQ)
Description: A self-report validated questionnaire to explore the child's perceptions of their asthma will be conducted at each study visit. Within and between group comparisons between groups will be explored. The B-IPQ has 8 items which are scored on a Likert scale 0-10 scoring system and an overall score is calculated. Minimum score is 0 and maximum score is 80. Overall score indicates degree in which illness is perceived threatening - higher scorer = more threatening view.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 26 [6 to 46] | 33 [12 to 49]
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 23.50 [9 to 55] | 26 [3 to 55]
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 21.00 [10 to 25] | 26 [2 to 47]

7. Secondary Outcome: Habit
Description: Measured by validated questionnaire the self-report behavioural automaticity index (SRBAI) to be conducted at each study visit. Within and between group comparisons between groups will be explored. The questionnaire has 4-questions which are rated on a Likert scale of strongly agree (1) - strongly disagree (5). An average of all 4 questions is calculated (minimum score 1, maximum score 5), 1 means no habit and 5 means strong habit.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline): number analyzed (Participants) | 16 | 15
  0-weeks (baseline) | 2.75 (1.09) | 2.91 (0.63)
  12-weeks: number analyzed (Participants) | 14 | 16
  12-weeks | 2.72 (0.57) | 2.50 (0.83)
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 2.69 (0.87) | 3.06 (0.69)

8. Secondary Outcome: Self-reported Adherence
Description: Measured by the validated Medication Adherence Report Scale for Asthma (MARS-A) questionnaire. Within and between group comparisons will be explored. Comparisons against EMD record of adherence will be explored. Questionnaire has 10 items on a scale of 1 = always to 5 = never Likert scale. An average of all items is calculated, minimum score 1 and maximum score 5. A score of 4.5 and above indicates high adherence.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 4.20 [2.9 to 4.7] | 4.1 [2.6 to 4.7]
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 4.30 [2.7 to 4.8] | 4.20 [3.00 to 4.90]
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 4.20 [3.20 to 4.90] | 4.10 [3.10 to 4.90]

9. Secondary Outcome: Change in Percentage ICS Adherence for Control Participants Between 12-weeks and 24-weeks
Description: Change in % ICS adherence for control group between 12-weeks and 24-weeks. Average % ICS adherence measured by EMD. EMD will electronically record date/time of asthma inhaler actuation. Data from EMD will be downloaded at study visit/s. Possible scores: 0% (poor adherence) to 100% (good adherence).
Time Frame: Change in % ICS adherence in control from study visit 2 (12-weeks) to study visit 3 (24-weeks)
Measure: Median (Full Range); unit: percentage of adherence
Groups:
- 12-weeks: % ICS adherence for control participants at 12-weeks
- 24-weeks: % ICS adherence for control participants at 24-weeks
Arm/Group | 12-weeks | 24-weeks
Number analyzed (Participants) | 13 | 12
percentage of adherence | 56 [7 to 87] | 31.5 [3 to 62]

10. Secondary Outcome: Change in Percentage ICS Adherence for Intervention Participants Between 12-weeks and 24-weeks
Description: Change in % ICS adherence for intervention group between 12-weeks and 24-weeks. Average % ICS adherence measured by EMD. EMD will electronically record date/time of asthma inhaler actuation. Data from EMD will be downloaded at study visit/s. Possible scores: 0% (poor adherence) to 100% (good adherence).
Time Frame: Change in % ICS adherence in intervention from study visit 2 (12-weeks) to study visit 3 (24-weeks)
Measure: Median (Full Range); unit: percentage of adherence
Groups:
- 12-weeks: % ICS adherence for intervention participants at 12-weeks
- 24-weeks: % ICS adherence for intervention participants at 24-weeks
Arm/Group | 12-weeks | 24-weeks
Number analyzed (Participants) | 11 | 8
percentage of adherence | 73 [23 to 89] | 39 [0 to 72]

11. Secondary Outcome: Comparison of Percentage ICS Adherence Between Groups at 24-weeks (Follow-up)
Description: Average % ICS adherence measured by EMD. EMD will electronically record date/time of asthma inhaler actuation. Data from EMD will be downloaded at study visit/s. Possible scores: 0% (poor adherence) to 100% (good adherence).
Time Frame: Comparison between groups at 24-weeks (follow-up)
Measure: Median (Full Range); unit: percentage of adherence
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 8 | 12
percentage of adherence | 31.5 [3 to 62] | 39 [0 to 72]

12. Secondary Outcome: Total Number of Asthma Attacks Over the Course of the Study
Description: Self-report measure of the number of asthma attacks from the start of the study (0-weeks) until end of study (24-weeks).
Time Frame: study visit 3 (24-weeks)
Measure: Number; unit: Number of attacks
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 12 | 13
Number of attacks | 1 | 3

13. Secondary Outcome: Incident Rate Ratio of Asthma Exacerbations
Description: Calculation of incident rate ratio of asthma exacerbations based upon self-report number of asthma attacks at study visit 2 and study visit 3 and total number of attacks at 24-weeks.
Time Frame: study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Self-reported number of asthma attacks collected was too low to calculate the incident rate ratio of asthma exacerbations.
Measure: Mean (Standard Deviation); unit: ratio (unitless number)
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 14 | 15
ratio (unitless number) | NA (NA) — Self-reported number of asthma attacks collected was too low to calculate the incident rate ratio of asthma exacerbations | NA (NA) — Self-reported number of asthma attacks collected was too low to calculate the incident rate ratio of asthma exacerbations

14. Secondary Outcome: Autonomous Motivation
Description: Measured by an adaptation of the Treatment Self-Regulation Questionnaire (TSRQ) for the purpose of this study. Within and between group comparisons will be explored. There are 4 items for autonomous motivation. All items are scores on a scale of 0 (not at all true) and 7 (very true). A total score is calculated from all 4 questions, minimum score 4 and maximum score 28. A higher score = higher motivation in either domain. Addition of 2 questions for intervention group only on a similar scoring scale (0 = not at all true - 7 = very true) about the influence of incentives over motivation which will be reported descriptively.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 22.50 [8 to 28] | 22.50 [13 to 28]
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 22 [12 to 27] | 20 [15 to 27]
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 26 [14 to 27] | 21 [6 to 27]

15. Secondary Outcome: Controlled Motivation
Description: Measured by an adaptation of the Treatment Self-Regulation Questionnaire (TSRQ) for the purpose of this study. Within and between group comparisons will be explored. There are 4 items for controlled motivation. All items are scores on a scale of 0 (not at all true) and 7 (very true). A total score is calculated from all 4 questions, minimum score 4 and maximum score 28. A higher score = higher motivation in either domain. Addition of 2 questions for intervention group only on a similar scoring scale (0 = not at all true - 7 = very true) about the influence of incentives over motivation which will be reported descriptively.
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 18.19 (5.39) | 16.81 (5.08)
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 14.73 (3.51) | 17.07 (4.73)
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 17.67 (5.16) | 15.38 (5.95)

16. Secondary Outcome: Belief in Medicine Questionnaire (BMQ) - Necessity
Description: A self-report validated questionnaire to explore the child's belief in their asthma medicines will be conducted at each study visit. Within and between group comparisons between groups will be explored. The questionnaire is split into 1) BMQ specific (medicines prescribed to child) that has 10 items and 2) BMQ - general (medicines in general) that has 8 items - all with a likert scale response of strongly agree - strongly disagree. Questions can be grouped into: necessity, concern, harm and over-use. Total scores for Necessity: 5 = low belief in need for medicine; 25 = high belief in need for medicine
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 15.19 (3.33) | 14.19 (3.25)
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 15.53 (2.89) | 16.21 (2.33)
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 16.17 (3.25) | 14.38 (3.25)

17. Secondary Outcome: Belief in Medicine Questionnaire (BMQ) - Concern
Description: A self-report validated questionnaire to explore the child's belief in their asthma medicines will be conducted at each study visit. Within and between group comparisons between groups will be explored. The questionnaire is split into 1) BMQ specific (medicines prescribed to child) that has 10 items and 2) BMQ - general (medicines in general) that has 8 items - all with a likert scale response of strongly agree - strongly disagree. Questions can be grouped into: necessity, concern, harm and over-use. Total score for concern: 5 = low belief in concern of medicine; 25 = high belief in concern of medicine
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 15.63 (2.33) | 14.31 (3.42)
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 15.33 (2.74) | 15.64 (2.53)
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 16.67 (3.34) | 15.31 (2.63)

18. Secondary Outcome: Belief in Medicine Questionnaire (BMQ) - Harm
Description: A self-report validated questionnaire to explore the child's belief in their asthma medicines will be conducted at each study visit. Within and between group comparisons between groups will be explored. The questionnaire is split into 1) BMQ specific (medicines prescribed to child) that has 10 items and 2) BMQ - general (medicines in general) that has 8 items - all with a likert scale response of strongly agree - strongly disagree. Questions can be grouped into: necessity, concern, harm and over-use. Total harm score: 4 = low belief in harm of medicine; 20 = high belief in harm of medicine
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 12.5 [6 to 17] | 12 [9 to 20]
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 14 [9 to 17] | 12 [10 to 17]
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 12.5 [7 to 18] | 13 [10 to 18]

19. Secondary Outcome: Belief in Medicine Questionnaire (BMQ) - Over-use
Description: A self-report validated questionnaire to explore the child's belief in their asthma medicines will be conducted at each study visit. Within and between group comparisons between groups will be explored. The questionnaire is split into 1) BMQ specific (medicines prescribed to child) that has 10 items and 2) BMQ - general (medicines in general) that has 8 items - all with a likert scale response of strongly agree - strongly disagree. Questions can be grouped into: necessity, concern, harm and over-use. Total over-use score: 4 = low belief in medicine over-use; 20 = high belief in medicine over-use
Time Frame: study visit 1 (0 weeks), study visit 2 (12-weeks) and study visit 3 (24-weeks)
Population: Participant numbers decrease between baseline, 12-weeks and 24-weeks due to participant withdrawal
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
Number analyzed (Participants) | 16 | 16
score on a scale
  0-weeks (baseline) | 15 [10 to 17] | 15 [10 to 18]
  12-weeks: number analyzed (Participants) | 14 | 15
  12-weeks | 15 [8 to 17] | 14 [10 to 16]
  24-weeks: number analyzed (Participants) | 12 | 13
  24-weeks | 15.5 [8 to 17] | 14 [10 to 18]

ADVERSE EVENTS:
Time Frame: Throughout study duration: 0-24-weeks
Description: It was unlikely any participants were at risk throughout this study as it was an interventional study using adherence monitoring and reminders (plus financial incentives for intervention participants)
Arm/Group | Control (no Financial Incentive) | Intervention (Financial Incentive)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 3/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (no Financial Incentive) (N=16) | Intervention (Financial Incentive) (N=16)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) — Number of asthma attacks were primarily data collected as an outcome measures for this study, but are also detailed here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT05322044/Prot_SAP_000.pdf